CLINICAL TRIAL: NCT01360788
Title: GOLD Stage I COPD: Is it Really a Disease ? Exercise Tolerance, Muscle Function and Response to Bronchodilation in GOLD Stage I COPD Patients
Brief Title: GOLD Stage I Chronic Obstructive Pulmonary Disease (COPD)
Acronym: GOLD
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Boehringer Ingelheim (Industry); Pfizer (Industry)
Responsible Party: Dr François Maltais, Institut Universitaire de cardiologie et de pneumologie de Québec
Other Study IDs: GOLD-20378
Record Dates: First submitted 2011-05-12; First posted 2011-05-26 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Mild Chronic Obstructive Pulmonary Disease; Respiratory Symptoms; Physical Activity
Keywords: chronic obstructive pulmonary disease; lung function; symptoms; activity-related dyspnea; quadriceps muscle function; exercise capacity; physical activity in daily life; muscle biopsy; systemic inflammation; GOLD stage I; pulmonary function
MeSH Terms: conditions — Signs and Symptoms, Respiratory; Motor Activity; Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Albuterol, Ipratropium Drug Combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Muscle biopsies Venous blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy control subjects: Subjects with a significant smoking history (more than 10 pack-years) and a normal lung function.
- Asymptomatic GOLD stage I COPD patients: GOLD stage I COPD (post-bronchodilator forced expiratory volume in 1 second [FEV1] > 80% predicted and FEV1/ forced vital capacity [FVC] < 0.7 and a smoking history > 10 pack-years) were recruited. A Medical Research Council (MRC) dyspnea score ≥ 2 was used to define the presence of symptoms (dyspnea). Concretely, this group did not present any respiratory symptoms, with a MRC dyspnea score of 1/5.
  Interventions: Drug: Combination ipratropium/salbutamol or placebo (nebulization)
- Symptomatic GOLD stage I COPD patients: GOLD stage I COPD (post-bronchodilator forced expiratory volume in 1 second [FEV1] > 80% predicted and FEV1/ forced vital capacity [FVC] < 0.7 and a smoking history > 10 pack-years) were recruited. A Medical Research Council (MRC) dyspnea score ≥ 2 was used to define the presence of symptoms (dyspnea) in this group.
  Interventions: Drug: Combination ipratropium/salbutamol or placebo (nebulization)

INTERVENTIONS:
Drug: Combination ipratropium/salbutamol or placebo (nebulization) — The COPD patients were randomly assigned a combination of ipratropium/salbutamol or a placebo in a double-blind crossover design. The bronchodilation produced by the medication was given in order to evaluate if bronchodilation was effective in increasing exercise tolerance during an endurance shuttle walking test in patients with GOLD stage I COPD.
  Other Names: Combivent or placebo (nebulization)
  Groups: Asymptomatic GOLD stage I COPD patients; Symptomatic GOLD stage I COPD patients

SUMMARY:
Recently integrated in clinical practice, the Global Initiative for Chronic Obstructive Lung Disease (GOLD) classification states that a mild (stage I) chronic obstructive pulmonary disease (COPD) is present, in a smoker, when the postbronchodilator forced expired volume in 1 second (FEV1) to forced vital capacity (FVC) ratio is < 0.7. A major change that was introduced by the GOLD classification system was that COPD could be diagnosed despite an FEV1 that is within normal predicted values (above 80% predicted). Because it suggests diagnosing and detecting COPD earlier than done until very recently in medical practice, the GOLD standards bring in a new reality to clinicians. In fact, this novel COPD classification comes with new research challenges because the functional impacts and systemic consequences related to COPD are mostly documented in patients with moderate to severe stages with little information specifically in GOLD stage I COPD. This information is important if the investigators are to convince physicians that GOLD stage I COPD needs to be diagnosed and eventually treated.

The investigators aimed to characterize GOLD stage I COPD patients according to activity-related dyspnea. More specifically, our objectives were to compare:

i) baseline pulmonary function ii) exercise capacity iii) quadriceps muscle function iv) levels of physical activity in daily life

between symptomatic (Sx) GOLD stage I COPD patients, asymptomatic (ASx) GOLD stage I COPD patients and healthy control subjects (CTRL). The investigators reasoned that exercise tolerance and physical activity levels would be decreased in Sx GOLD stage I COPD patients as it would be similar between ASx GOLD stage I COPD patients and CTRL.

DETAILED DESCRIPTION:
The study will be conducted among three subgroups: symptomatic GOLD stage I patients with COPD, asymptomatic patients GOLD stage I COPD and healthy control subjects with normal lung function. Subjects will be paired for age, sex and smoking history. The project will require three visits. In the initial visit, assessment of the pulmonary function with respiratory symptoms quantification will allow to classify subjects in the proper subgroup. The Medical Research Council (MRC) dyspnea scale will serve as the reference outcome to determine whether COPD patients are symptomatic or not. Patients with an MRC dyspnea score < 2 will be considered asymptomatic. A second questionnaire (ATS-DLD-78) will serve to document cough, expectorations, wheezing and smoking history in every subjects. Body composition will be measured by bioimpedance and by waist circumference after a blood sample taken in the morning, in a fasting state. A six-minute walk test (6MWT) will be performed by all subjects. After a one-hour resting period, a maximal incremental shuttle walking test will be realized in the same visit to quantify maximal exercise capacity. Measures of force and endurance of the quadriceps will be taken by magnetic stimulation of the femoral nerve before the maximal walking test. Finally, subjects will receive a portable device to monitor physical activity for a period of 7 days.

In the 2nd and 3rd visits, subjects will realize an endurance walking test at 85 % of their predetermined maximal capacity. Before each endurance test, a bronchodilator or a placebo will be administered following a randomized double-blind design. Measures of force and endurance of the quadriceps will be taken by magnetic stimulation of the femoral nerve before and 10-min after endurance exercise tests. A needle biopsy of the vastus lateralis will be performed at the end of the third visit.

ELIGIBILITY:
Inclusion Criteria:

* Smoking history (≥ 10 pack/year)

Exclusion Criteria:

* Anticoagulation or coagulation defect
* Hypoxemia or exercise-induced desaturation (SpO2 < 85%)
* Antibiotic or oral corticosteroid therapy (end of treatment < 1 month prior to study)
* Anti-inflammatory treatment, exacerbation (< 3 months)
* Myopathy
* Neuromuscular or locomotor diseases
* Recent cancer
* Unstable cardiac condition
* Asthma

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were recruted after a participation to a research protocol on i) prevalence of COPD in Canada and ii) early detection of lung cancer. Finally, some participants were recruited following medical consultation with a pneumologist.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2009-02; Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption | Baseline
  Exercise capacity was directly assessed following an incremental progressive shuttle test. The exercise capacity was defined as the maximal oxygen consumption (VO2 peak, ml/kg/min) by direct measurements of gas exchanges.

SECONDARY OUTCOMES:
Quadriceps muscle force | Baseline
  Quadriceps muscle strength was measured with magnetic stimulation of the femoral nerve.
  Mid-thigh cross-sectional area (MTCSA) was obtained following a computed-tomography scan.
  Quadriceps muscle biopsy was performed to measure muscle metabolism.
Levels of physical activity in daily life | Baseline
  A portable armband was worn by the participants on a 7-days basis to monitor physical activities in daily life.
Oxydative stress | Baseline
  Oxydative stress will be quantified in the blood and in the muscle samples obtained during the muscular biopsy.
Pulmonary function | At baseline and before and 60-min after the nebulization of either placebo or bronchodilator
  Pulmonary function will be measured by spirometry and plethysmography in the initial visit. In the subsequent visits, pulmonary function will be measured by spirometry before and 60-min after the nebulization of either placebo or bronchodilator. A computed-tomography scan of the lungs was also assessed
Time to exhaustion during a constant intensity exercise test | Before and 90-min after bronchodilation or placebo
  Time to exhaustion was also defined as exercise tolerance and was assessed during a endurance shuttle walking test 90-min following the nebulization of whether Combivent or Placebo in a double-blind crossover design. It was defined as the time in seconds for which a subject could maintain an intensity of 85% of the maximal oxygen consumption during walking or running.
Systemic inflammation | Baseline
  Systemic inflammation will be studied from blood samples obtained in every participants.
Quadriceps muscle endurance | Baseline
  Quadriceps muscle endurance was defined as the time to exhaustion following a constant quadriceps force corresponding to 50 % of the maximal voluntary contraction.

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Gagnon P, Casaburi R, Saey D, Porszasz J, Provencher S, Milot J, Bourbeau J, O'Donnell DE, Maltais F. Cluster Analysis in Patients with GOLD 1 Chronic Obstructive Pulmonary Disease. PLoS One. 2015 Apr 23;10(4):e0123626. doi: 10.1371/journal.pone.0123626. eCollection 2015. PMID 25906326